CLINICAL TRIAL: NCT04101227
Title: Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy, Safety and Tolerability of AD04 (Ondansetron) in Adults With Alcohol Use Disorder (AUD) and Selected Polymorphisms in the Serotonin Transporter and Receptor Genes
Brief Title: Study to Evaluate AD04 in Adults With Alcohol Use Disorder (AUD) and Selected Serotonin Transporter Polymorphisms
Acronym: ONWARD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Adial Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AD04-301
Record Dates: First submitted 2019-09-23; First posted 2019-09-24 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Ondansetron; Genetic Testing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment Arm (Experimental): AD04 (ondansetron)
  Interventions: Drug: AD04 (ondansetron); Device: Companion Diagnostic for Genetic Testing; Behavioral: Brief Psychological Counseling
- Placebo Arm (Placebo Comparator): Matching Placebo
  Interventions: Drug: Matching placebo; Device: Companion Diagnostic for Genetic Testing; Behavioral: Brief Psychological Counseling

INTERVENTIONS:
Drug: AD04 (ondansetron) — AD04 (ondansetron) 0.33 mg, orally (p.o.) twice a day (BID)
  Arms: Treatment Arm
Drug: Matching placebo — Matching placebo to AD04 (ondansetron), orally (p.o.) twice a day (BID)
  Arms: Placebo Arm
Device: Companion Diagnostic for Genetic Testing — Companion Diagnostic for Genetic Testing
Behavioral: Brief Psychological Counseling — Brief Psychological Counseling

SUMMARY:
Randomized, multi-center, double-blind, parallel-group, placebo-controlled study. Eligible subjects will be randomized to receive either 0.33 mg AD04 or placebo orally twice-daily for 24 weeks in conjunction with brief psychological counseling. Randomization will be stratified by:

1. Level of alcohol consumption prior to enrollment in the study (heavy drinkers averaging <10 drinks per day of drinking or very heavy drinkers averaging ≥10 drinks per day of drinking), and
2. Gender (male or female).

DETAILED DESCRIPTION:
Target enrollment of subjects with AUD who regularly engage in risk alcohol consumption (i.e. >6/day or more heavy alcohol consumption in the 4 weeks preceding the screening visit), and have selected genotypes (LL/TT genotype and/or 1, 2 or 3 of the SNPs on the genes for the 5-HT3 receptor subunits: rs1150226-AG or rs1176713-GG in the gene that encodes the 5-HT3A receptor subunit, and rs17614942-AC in the gene that encodes the 5-HT3B receptor subunit), and who are eligible to participate in the study based on meeting the remaining study inclusion/exclusion criteria. Eligible subjects will be randomized to receive either 0.33 mg AD04 or placebo BID for 24 weeks.

The trial will have a 16-week grace period to enable medication effects to be optimal for comparison with placebo. The grace period starts immediately after beginning of study drug treatment, in which consumption of alcohol is not counted as a failure. All primary and secondary efficacy endpoints will be assessed during the last 8 weeks of treatment (i.e. weeks 17-24). The primary measure of efficacy, incidence risk alcohol consumption, will be assessed over the last 8 weeks of treatment. The secondary measure of efficacy evaluating the incidence of risk alcohol consumption over the last 4 weeks of treatment, important because it has been used commonly to validate efficacy for regulatory agencies such as the European Medicines Agency, was also calculated. To enhance study feasibility, subjects will be evaluated every week during the first 8 weeks of treatment and every other week for the remaining 16 weeks of the treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. The subject has signed the Informed Consent Form.
2. The subject has breath alcohol concentration (BAC) of 0.00% at the Screening and < 0.02 % at the Baseline visit.
3. The subject has moderate to severe diagnosis of AUD as measured by Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria.
4. Males and females aged 18 and over.
5. Able to provide Timeline Follow-back Method (TLFB) alcohol consumption information for the 28-day period prior to Screening Visit.
6. A subject is eligible for participation in the study if he/she had:

   1. ≥6 HDDs (HDD is defined as a day with alcohol consumption of 60 g or more for males and 40 g or more for females) in the 4 weeks prior to the Baseline Visit,
   2. an average alcohol consumption at the medium risk level (defined by the WHO "International guide for monitoring alcohol consumption and related harm" as >40 grams of ethanol/day for males and >20 grams of ethanol/day for females) for the 4 weeks prior to the Screening Visit,
   3. ≤14 consecutive abstinent days in the 4 weeks preceding the Screening Visit.
7. Willingness to provide a blood sample for DNA analysis at the Screening visit. The blood sample collected for DNA testing contains at least one of the following genotypes as measured by Adial's validated method:

   * rs4795541-LL genotype of the insertion-deletion polymorphism (5'-HTTLPR) in the 5'-regulatory region and rs1042173-TT SNP in the 3'-untranslated region of SLC6A4 gene that encodes the serotonin transporter
   * rs1150226-AG SNP in HTR3A, the gene that encodes subtype A of the serotonin-3 receptor
   * rs1176713-GG SNP in HTR3A, the gene that encodes subtype A of the serotonin-3 receptor
   * rs17614942-AC in HTR3B, the gene that encodes subtype B of the serotonin-3 receptor
8. Expressed a wish to reduce or stop alcohol consumption.
9. Willingness to participate in behavioral and medicinal treatments for AUD.
10. Has had a stable residence in the 28 days prior to the Baseline Visit in the study and has no plans to move in the next 9 months. A stable residence is a domicile in which an individual can operate as if it were his or her own homestead and does not include shelters or halfway houses.
11. Provides contact information for 2 individuals who can be used to contact the subject.
12. Able to read and understand, and complete the rating scales and questionnaires accurately, follow instructions, and make use of the behavioral treatments.
13. The subject, if female must:

    * have a negative urine pregnancy test prior to the initiation of treatment and agree not to try to become pregnant during the study
    * use two adequate methods of contraception [intrauterine device, oral contraceptives, progesterone implanted rods, or regular medroxyprogesterone acetate injections in addition to condom or diaphragm, or double barrier method (condom or diaphragm + spermicide)], or
    * be post-menopausal having had the last natural menstruation at least 24 months prior to the Screening Visit, or
    * have had a hysterectomy or been surgically sterilized prior to baseline.

Exclusion Criteria:

1. Patients with withdrawal symptoms requiring additional medication for withdrawal. If present at Screening/Baseline Visit, subjects must complete a medically supervised detoxification program prior to being able to enroll in the study.
2. Subjects with diagnosis of any of the following concomitant psychiatric disorders: non-treated, unstable schizophrenia, bipolar disorder, other psychotic disorder during the lifetime of the subject. Recent (within last 12 months) diagnosis of a major depressive disorder, post traumatic stress disorder, panic disorder or eating disorders. Subjects with nicotine use disorder, phobic or other anxiety disorders (other than post-traumatic stress disorder or panic disorder) can be included.
3. The subject reports current or recent (within 8 weeks prior to Baseline Visit) treatment with antipsychotics or antidepressants medications, which can have an effect on serotonin receptor or transporter actions.
4. The subject has been treated with any investigational medicinal product within 30 days or 5 half-lives (whichever is longer) prior to the Baseline Visit.
5. The subject is currently participating or has recently (4 weeks prior to the Baseline Visit) participated in a treatment program for alcohol use disorders.
6. Any subject who has suicidal thoughts as evaluated by the Columbia Suicide Severity Rating Scale (C-SSRS) (i.e., has any suicidal ideation of type 4 or 5 on the C-SSRS in the last month).
7. The subject has a clinically significant untreated and unstable illness, for example, hepatic or renal insufficiency, or a cardiovascular, pulmonary, gastrointestinal, endocrine, neurological, infectious, neoplastic, or metabolic disturbance.
8. The subject has clinically significant abnormal vital signs.
9. The subject has a clinically abnormal ECG at the Screening/Baseline Visit, clinically significant cardiovascular disease requiring regular or intensive clinical monitoring, a current history of arrhythmias, or a current or past history of clinically significant QT prolongation, including:

   * QTcF > 450 ms (one ECG at screening and average of 3 12-lead measurements at baseline)
   * serum potassium, magnesium or calcium levels outside the central laboratory's reference range
   * receiving medications (within the last 7 days prior to the Baseline Visit) that have the potential of prolonging the QT interval or may require such medications during the course of the study
   * clinically unstable cardiac disease, including unstable atrial fibrillation, symptomatic bradycardia, unstable congestive heart failure, active myocardial ischemia or indwelling pacemaker
   * complete left bundle branch block
   * history of Long QT Syndrome or an immediate family member with this condition
10. The subject with elevated liver function tests or diagnosis of hepatic failure, esophageal variceal disease or any other clinically significant hepatic disease. The clinical evidence may include any of the following: prolonged prothrombin time (International Normalized Ratio, INR≥1.7) with bilirubin > 10% above the upper limit, and/or serum glutamic oxaloacetic transaminase (SGOT), and/or serum glutamic pyruvic transaminase (SGPT) and/or lactate dehydrogenase (LDH) > 3x the upper limit of normal at screening.
11. The subject reports treatment, either current or within 28 days prior to the Baseline Visit, with any medications having a potential effect on alcohol consumption and related behaviors or mood. These include opiate antagonists (e.g., naltrexone, Vivitrol®, Selincro®), glutamate antagonists (e.g., acamprosate), anticonvulsants (e.g., topiramate), serotonin reuptake inhibitors (e.g., fluoxetine), serotonin antagonists (e.g., buspirone), other antidepressants (e.g., tricyclic antidepressants or monoamine oxidase inhibitors), dopamine antagonists (e.g., haloperidol), and disulfiram (Antabuse®). Note benzodiazepines are allowed if used chronically.
12. Previous or current abuse of benzodiazepines.
13. At Baseline Visit, the subject's urine contains prescription and non-prescription drugs with abuse potential or other psychotropic agents not otherwise specified, including herbal agents such as St John's Wort that could interfere with the drug treatment.
14. The subject has a history of allergic reactions or other known intolerance to ondansetron or other 5-HT3 antagonists.
15. Female subjects of childbearing potential who have a positive pregnancy test at Screening/Baseline Visit or are pregnant, breast feeding and who are unwilling to adhere to an acceptable form of contraception or meet the other criteria for inclusion as specified for females in the inclusion criteria (See Inclusion Criteria, Item # 13).
16. The subject received in-patient or out-patient treatment for alcohol use disorder within the 28 days prior to the Baseline Visit.
17. As of the Baseline Visit, the subject is compelled to participate in an alcohol treatment program to maintain his/her liberty.
18. As of Baseline Visit, the subject is sharing a household with a subject randomized to any investigational trial of ondansetron.
19. Any other condition or therapy that in the investigator's opinion may pose a risk to the subject, prevent the subject from completing the required study procedures or interfere with the study objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-03-18 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the percentage of monthly heavy drinking days (PHDD) | Weeks 16 to 24
  Change from baseline in the percentage of monthly HDDs, where (heavy) drinking is defined as the consumption of ≥ 60 g alcohol/day (if male) or ≥ 40 g alcohol/day (if female).

SECONDARY OUTCOMES:
Change from baseline in the primary efficacy endpoint at each study month | Weeks 4, 8, 12, 16, 20, and 24
  Change from baseline in PHDD at each study month.
Change from baseline in AUD symptoms and clinical status | Weeks 12 and 24
  AUD symptoms and clinical status (<2 symptoms, Mild, Moderate, or Severe) based on DSM-5 criteria at Baseline, weeks 12 and 24 visits
Change from baseline in Drinking Risk Levels (DRL), 1-level shift | Week 24
  Proportion of subjects with a 1-level categorical shift from baseline in modified DRL
Change from baseline in Drinking Risk Levels (DRL), 2-level shift | Week 24
  Proportion of subjects with a 2-level categorical shift from baseline in modified DRL
Change from baseline in total alcohol consumption (TAC) | Weeks 16 to 24
  Change from baseline in total alcohol consumption (TAC), defined as the mean daily alcohol consumption expressed in g/day
Change from baseline in the Patient Health Questionnaire-9 (PHQ-9) | Week 24
  Change from baseline in the PHQ-9 calculated as the difference from baseline to Week 24.
Change from baseline in risk alcohol consumption responders | Weeks 16 to 24
  The number of subjects with no risk alcohol consumption will be calculated
Change from baseline in percent reduction in monthly total alcohol consumption (TAC) | Weeks 20 to 24
  Proportion of subjects with ≥10%, ≥20%, ≥30%, ≥40%, ≥50%, ≥60%, ≥70%, ≥80%, and ≥90% reduction from baseline in monthly TAC
Change from baseline in the percent of non-drinking days (PNDD) | Weeks 16 to 24
  Change from baseline in the percent of non-drinking days (PNDD)
Change from baseline in drinks per drinking day (DDD) | Weeks 16 to 24
  Change from baseline in the monthly drinks per drinking day (DDD)

CONTACTS AND LOCATIONS:
Overall Officials: Professor, Dr Hannu Alho, Principal Investigator — National Institute for Health and Welfare Research Center Biomedicum
Locations (25):
- Bulgaria (7):
  - Mental Health Centre Prof. Dr. Ivan Temkov Burgas EOOD Department for treatment of Emergency Psychiatric conditions, Burgas
  - State Psychiatric Hospital, Kardzhali
  - UMHAT Dr. Georgi Stranski Second Psychiatric Clinic, Pleven
  - Ambulatory for Group Practice for Specialized Psychiatric Help - Philipopolis OOD, Plovdiv
  - Medical Center Intermedica OOD, Sofia
  - State Psychiatric Hospital for Treatment of drug addiction and alcoholism, Sofia
  - Diagnostic-Consultative Center Mladost-М Varna, Varna
- Croatia (3):
  - Clinical Hospital Center Split, Split
  - Polyclinic Neuron, Zagreb
  - University Psychiatric Hospital Vrapče Klinika za psihijatriju Vrapče, Zagreb
- West Tallinn Central Hospital, Haabersti Health Center, Tallinn, Estonia
- Finland (6):
  - Addiktum klinikka Helsinki, Helsinki
  - Savon psykiatripalvelu, Kuopio
  - Mentalcare, Oulu
  - Satakunnan Psykiatripalvelu Oy, Pori
  - Satakunnan Psykiatripalvelu Oy, Tampere
  - Addiktum Oy, Turku
- Latvia (3):
  - Liepaja Regional Hospital Addictive disorder department, Liepāja
  - M&M Centrs, Riga
  - Strenci Psychoneurological Hospital, Strenči
- Poland (3):
  - Centrum Medyczne Luxmed Sp. z. o. o., Lublin
  - NZOZ Prywatna Klinika Psychiatryczna, Tuszyn
  - Clinical Research Group Sp. z.o.o, Warsaw
- Sweden (2):
  - Ladulaas Kliniska Studier, Borås
  - ClinSmart Sweden AB, Uppsala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Prospective Pharmacogenetic Phase 3 Clinical Trial of Low-Dose Ondansetron (A 5-HT3 Antagonist) to Treat Heavy and Very Heavy Drinkers With Alcohol Use Disorder — https://doi.org/10.21203/rs.3.rs-2156237/v1
- See also: Safety and compliance of long-term low-dose ondansetron in alcohol use disorder treatment — https://linkinghub.elsevier.com/retrieve/pii/S0953-6205(24)00123-7